CLINICAL TRIAL: NCT02721953
Title: Effects of Butyrate on Insulin Resistance in Children Affected by Obesity
Brief Title: The Effects of Butyrate on Children With Obesity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29/14
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypocaloric diet plus butyrate (Experimental): Hypocaloric diet plus butyrate
  Interventions: Dietary Supplement: Butyrate
- Hypocaloric diet plus placebo (Placebo Comparator): Hypocaloric diet plus placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Butyrate — Butyrate
  Arms: Hypocaloric diet plus butyrate
Other: Placebo — Placebo
  Arms: Hypocaloric diet plus placebo

SUMMARY:
Butyrate is a short chain fatty acid (SCFA) produced by bacterial fermentation of undigested starch in the gut. Butyrate carries out different effects at intestinal and extraintestinal level, including: immune regulation with anti-inflammatory effect at intestinal and systemic level and modulation of gut microbiota. Many of these effects result from an epigenetic mechanism. Shown in an animal model of obesity induced by a high fat diet (HFD), that butyrate can exercise very effective protective action against obesity through the stimulation of intestinal satiety hormones. Shown always in murine model of obesity induced by HFD, that butyrate is effective in preventing and treating obesity and insulin resistance. After 5 weeks of treatment with butyrate was observed a reduction of 10.2% of body weight, 30% of fasting glucose and 50% insulin resistance.

In an animal model of metabolic syndrome with NAFLD researchers have recently demonstrated that the administration of butyrate is able to significantly reduce insulin resistance, liver damage, dyslipidaemia through a modulation of the inflammatory process.

Pharmacokinetic and pharmacodynamic studies in humans show that the oral administration of butyrate is safe and well tolerated. The peak serum levels occurs 4-6 hours after oral administration.

All of these data makes plausible a possible positive effect on insulin resistance in the obese child.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI >95° percentile)
* HOmeostasis Model Assessment (HOMA-IR) > 4 (obtained by calculating the product of fasting plasma insulin expressed in microunits/mL and fasting plasma glucose expressed in mmol/L divided by 22.5)

Exclusion Criteria:

* Age <10 or >15 years
* BMI <95° centile
* HOMA-IR <4
* Patients under pharmacological treatment for obesity (metformin) or taking vitamin E, pre-, pro- or synbiotics
* Simultaneous presence of other chronic diseases unrelated to obesity (cancer, immunodeficiency, cystic fibrosis, allergies, celiac disease, autoimmune diseases, neuropsychiatric disorders, type 1 diabetes, inflammatory bowel diseases, malformations of urinary or gastrointestinal or respiratory tract, chronic lung diseases, genetic and metabolic diseases, chronic hematological diseases)
* History of surgery for the treatment of obesity
* Any medical condition that may interfere with participation in this study
* Participation in other clinical trials still in progress

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of insulin resistance | After 6 months of treatment

SECONDARY OUTCOMES:
Reduction of body weight | After 6 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No